CLINICAL TRIAL: NCT03655561
Title: Observational Cohort Study of Lassa Fever Clinical Course and Prognostic Factors in an Epidemic Context in Nigeria
Brief Title: Lassa Fever Clinical Course and Prognostic Factors in Nigeria
Acronym: LASCOPE
Status: Active, not recruiting | Type: Observational
Sponsor: Alliance for International Medical Action (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); University of Oxford (Other); Irrua Specialist Teaching Hospital (Other); Bernhard Nocht Institute for Tropical Medicine (Other Government); University Hospital, Bordeaux (Other); University of Bordeaux (Other); PACCI Program (Other); Institut de Recherche pour le Developpement (Other Government); ANRS, Emerging Infectious Diseases (Other Government); Federal Medical Centre, Owo (Industry); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Principal Investigator, Denis Malvy, Professor of Infectious Diseases and Tropical Medicine, Alliance for International Medical Action
Other Study IDs: LAS001
Record Dates: First submitted 2018-08-30; First posted 2018-08-31 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Lassa Fever; Lassa Virus Infection; Pregnancy Complications; Acute Kidney Injury; Acute Kidney Failure; Coma
Keywords: Lassa fever; Lassa virus; Nigeria; Pregnancy; Acute kidney injury
MeSH Terms: conditions — Lassa Fever; Pregnancy Complications; Acute Kidney Injury; Coma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Days
Biospecimen Retention: Samples With DNA — Leftover blood, urine, milk and any other bodily fluid samples. Option for genetic analyses regarding immunity against infectious diseases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Confirmed Lassa fever cases: Participants with a clinical presentation consistent with acute Lassa virus disease and a positive result for Lassa specific RT-PCR obtained before or after inclusion
  Interventions: Other: Non interventional research
- Non-Lassa cases (controls): Participants with a clinical presentation consistent with acute Lassa virus disease but subsequently found to have a negative result for Lassa specific RT-PCR
  Interventions: Other: Non interventional research

INTERVENTIONS:
Other: Non interventional research — Participants are receiving the standard of care according to Nigerian Center for Disease Control (NCDC) Standard Operating Procedures for Lassa fever case management. This include the administration of intravenous ribavirin for Lassa confirmed cases as well as critically-ill Lassa suspected cases.

SUMMARY:
The investigators propose to conduct a nationwide (Nigeria), prospective, non-interventional cohort study describing the clinical course, biological characteristics, case management and outcomes in patients hospitalized for a suspected or confirmed diagnosis of Lassa fever in tertiary medical facilities situated in the most affected Nigerian states. Special focuses will be made on situations at risk of bad outcome such as pregnancies, acute kidney injury and electrolytic imbalance in patients with confirmed Lassa fever. Participants for which the diagnosis of Lassa fever will be finally excluded by reverse-transcriptase polymerase chain reaction (RT-PCR) will constitute the control group.

DETAILED DESCRIPTION:
The LASCOPE project refers to a nationwide, prospective, non-interventional cohort study describing the clinical course, biological characteristics, case management and outcomes in patients hospitalized for a suspected or already RT-PCR confirmed diagnosis of Lassa fever in tertiary medical facilities situated in the most affected Nigerian states. The project will start during the 2018 Lassa fever season and is intended to be extended to at least three sites throughout Nigeria on a 3 years period.

The investigators will try to depict the pathophysiological mechanisms underlying the conditions associated to a fatal outcome in patients with RT-PCR confirmed Lassa fever, with a special focus on pregnancies, acute renal injury and electrolytic imbalance.

Population and setting - Participants will be recruited in tertiary reference hospitals for Lassa fever case management in the Nigerian States identified to have the highest burden, including Owo Federal Medical Center (OFMC), Owo, Ondo State as a pilot site (list to be completed according to the outbreak dynamics).

Inclusion criteria - All the patients hospitalized for suspected or already RT-PCR confirmed Lassa fever will be eligible (no age restriction). Newborns from mothers participating in the study will also be eligible.

Sample size - Given the descriptive purpose of the study, there is no pre-determined sample size.

Follow-up - After informed consent collection, data concerning the patient's life habits, contacts, disease history, clinical and biological status, management and outcome will be collected anonymously upon admission and throughout the hospital stay. The follow-up will end 60 days after admission (60 days after delivery for pregnant women and 60 days after birth for newborns) with a phone call or a home visit (or an outpatient visit at hospital if needed).

Leftover biological samples, if any, will be stored for further analysis with the participant's agreement. The biobank will be registered once constituted and further use of stored samples will be subject to material transfer agreements.

ELIGIBILITY:
Inclusion Criteria:

* EITHER admission (inpatient) for suspected or already RT-PCR confirmed Lassa fever OR newborn from woman infected with Lassa virus during pregnancy
* AND written informed consent of the patient or his/her legal representative (specific procedures for: immature minors, mature minors, incapable adults and unconscious adults; witnessed consent in case of illiteracy)

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients admitted in an isolation ward of one of the participating sites (tertiary hospitals) in Nigeria for a suspected or already RT-PCR confirmed diagnosis of Lassa fever during the study period are eligible to participate in LASCOPE.
  The newborns from women infected by Lassa virus (RT-PCR confirmed) during their pregnancy are also eligible to participate, with the mother's agreement.
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2018-04-05 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall mortality | 60 days after admission (day 60 after delivery for pregnant women and day 60 after birth for newborns from infected pregnant women).
  Mortality rate among participants assessed at final visit.

SECONDARY OUTCOMES:
Acute kidney injury | Within 60 days after admission
  Acute kidney injury or failure according to RIFLE criteria
Mother status at the end of pregnancy | Delivery
  Is the mother dead or alive at the end of pregnancy
Type of pregnancy termination | Delivery
  Spontaneous delivery, induced delivery, cesarean section, medical interruption, miscarriage
Pregnancy complications | Delivery
  Reporting any type of pregnancy complications
Newborn status at birth | Birth
  Is the newborn dead or alive
Newborn status at day 30 | Day 30 after birth
  Is the newborn dead or alive
Newborn status at day 60 | Day 60 after birth
  Is the newborn dead or alive

CONTACTS AND LOCATIONS:
Overall Officials: Denis Malvy, MD, PhD, Principal Investigator — Inserm 1219 - Infectious Diseases in Ressource Limited Countries; Oladele O Ayodeji, MD, Principal Investigator — Owo Federal Medical Centre
Locations (2):
- Nigeria (2):
  - Alex Ekwueme Federal University Teaching Hospital Abakaliki, Abakaliki, Ebonyi State
  - Owo Federal Medical Centre (Owo FMC), Owo, Ondo State

IPD SHARING:
Plan to Share IPD: Yes
IPD underlying results in scientific publications will be made available through the deposition of a datafile in a public data repository.
Supporting Information: Study Protocol
Time Frame: Upon publication of related scientific works (undefined duration).
Access Criteria: Free access.

REFERENCES:
- [Derived] Duvignaud A, Jaspard M, Etafo IC, Serra B, Abejegah C, Gabillard D, Doutchi M, Alabi JF, Adedokun MA, Akinpelu AO, Oyegunle OO, Etafo J, Dede AO, Onyechi MN, Ireneh MU, Gbenga-Ayeni O, Fadiminiyi KG, Ehigbor PI, Ouattara E, Levy-Marchal C, Karcher S, N'guessan-Koffi L, Ahyi I, Amani E, Diabate M, Siloue B, Schaeffer J, Augier A, Ogbaini-Emovon E, Salam AP, Horby P, Ahmed LA, Gunther S, Adedosu AN, Anglaret X, Ayodeji OO, Malvy D. Lassa fever clinical course and setting a standard of care for future randomized trials: A protocol for a cohort study of Lassa-infected patients in Nigeria (LASCOPE). Travel Med Infect Dis. 2020 Jul-Aug;36:101557. doi: 10.1016/j.tmaid.2020.101557. Epub 2020 Jan 21. PMID 31978611